CLINICAL TRIAL: NCT06701396
Title: A Double-Blind, Randomized, Two-Period Crossover Study to Evaluate the Effects of Tasimelteon Vs. Placebo in Subjects with Delayed Sleep-Wake Phase Disorder (DSWPD) and the CRY1Δ11 Variant
Brief Title: Evaluating the Effects of Tasimelteon Vs. Placebo in Delayed Sleep-Wake Phase Disorder (DSWPD) and the CRY1Δ11 Variant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3501
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Chronobiology Disorders; Gene Mutations and Other Alterations Nec
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm; Chronobiology Disorders | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tasimelteon (Experimental)
  Interventions: Drug: Tasimelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasimelteon — Oral capsule
  Arms: Tasimelteon
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, two-period crossover study to evaluate the efficacy and safety of a single oral dose of tasimelteon and matching placebo in male and female subjects with DSWPD and the CRY1Δ11 variant.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent.
* A confirmed clinical diagnosis of Delayed Sleep-Wake Phase Disorder (DSWPD).
* Carrier of CRY1Δ11 variant.
* Men or women between 18 - 75 years, inclusive.
* Body Mass Index (BMI) of ≥ 18 and ≤ 40 kg/m^2.

Exclusion Criteria:

* Major surgery, trauma, illness, general anesthesia, or immobility for 3 or more days within the last 30 days.
* Pregnancy, recent pregnancy (within 6 weeks), or women who are breastfeeding.
* A positive test for substances of abuse.
* Current tobacco user.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Latency to Persistent Sleep, as measured by polysomnography. | Two Nights

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No